CLINICAL TRIAL: NCT05451160
Title: A Multicenter, Randomized, Parallel-controlled Clinical Trial Protocol to Validate the Safety and Efficacy of a Steep Pulse Therapy System for the Treatment of Liver Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Zhejiang Cancer Hospital (Other); West China Hospital (Other); Tianjin Third Central Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: steeppulse001
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-06

CONDITIONS: A Steep Pulse Therapy System for the Treatment of Liver Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steep Pulse Therapy System (Experimental)
  Interventions: Device: steep pulse therapy system
- RF Ablation System (Active Comparator)
  Interventions: Device: RF Ablation System

INTERVENTIONS:
Device: steep pulse therapy system — The steep pulse therapy system is produced by Zhejiang CuraWay Medical Technology Co., Ltd. for liver tumor ablation
  Arms: Steep Pulse Therapy System
Device: RF Ablation System — RF Ablation System
  Arms: RF Ablation System

SUMMARY:
This clinical trial is a multicenter, randomized, parallel-controlled study. In this study, patients with liver cancer were selected as the research subjects, and the subjects were randomly divided into the experimental group and the control group. The experimental group used the steep pulse treatment system produced by Zhejiang CuraWay Medical Technology Co., Ltd., and the control group used the RF Ablation System produced by Covidien llc. A total of 5 or 9 visits were planned in this study, namely the screening period (-14-0 days), the day of the first ablation, 2 ± 1 days after the first ablation, 30 ± 5 days after the first ablation, and after the first ablation 90±7 days, the day of secondary ablation, 2±1 days after secondary ablation, 30±5 days after secondary ablation, and 90±7 days after secondary ablation. The complete ablation rate at 30 ± 5 days after the first ablation was used as the main efficacy evaluation index to evaluate the safety and efficacy of the steep pulse therapy system produced by Zhejiang CuraWay Medical Technology Co., Ltd. for liver tumor ablation.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the patient is between 18-80 years old, and the gender is not limited.
2. For clinically diagnosed liver tumors, the diameter of a single tumor is less than or equal to 5cm; for multiple tumors: the number of tumors is not more than 3, and the largest tumor diameter is less than or equal to 3cm.
3. Patient is able to take care of himself, and ECOG performance status is between 0 and 2 points.
4. Liver function classification Child-Pugh A or B.
5. Expected survival period ≥ 6 months.
6. Patient is able to understand and comply with the trial protocol, and sign the informed consent.

Exclusion Criteria:

1. It is less than 30 days after the end of chemotherapy, radiotherapy, immunotherapy, or targeted therapy.
2. Within 3 months after ablation, patients need to continue treatment with chemotherapy, radiation therapy, immunotherapy, targeted therapy, surgery, or other minimally invasive modalities.
3. patients with severe infectious diseases such as bacteremia and toxemia.
4. patients with uncorrectable coagulation dysfunction (PLT<40xl09/L).
5. patients with severe heart, brain, lung and other diseases, and patients with severe arrhythmia.
6. patients with implanted artificial hearts, lungs, internal pulse regulators or wearable medical electronic devices such as electrocardiography.
7. Patients with a history of epilepsy.
8. Patients with acute myocardial infarction within 6 months.
9. Pregnant and lactating women and those who plan to become pregnant within one year.
10. Those who are allergic to ultrasound, CT or MRI contrast agents.
11. Those who are contraindicated in general anesthesia.
12. Those who have participated in clinical trials of any drug or medical device within the first 3 months of the group.
13. The researchers believe that there are other factors that are not suitable for inclusion or that affect the participation of subjects in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day complete ablation rate | 30 days
  Complete ablation rate

SECONDARY OUTCOMES:
Total complete ablation rate | 90 days
Success rate of puncture | 1 day
Equipment failure rate | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meijerink MR, Ruarus AH, Vroomen LGPH, Puijk RS, Geboers B, Nieuwenhuizen S, van den Bemd BAT, Nielsen K, de Vries JJJ, van Lienden KP, Lissenberg-Witte BI, van den Tol MP, Scheffer HJ. Irreversible Electroporation to Treat Unresectable Colorectal Liver Metastases (COLDFIRE-2): A Phase II, Two-Center, Single-Arm Clinical Trial. Radiology. 2021 May;299(2):470-480. doi: 10.1148/radiol.2021203089. Epub 2021 Mar 16. PMID 33724066
- [Result] Su GL, Altayar O, O'Shea R, Shah R, Estfan B, Wenzell C, Sultan S, Falck-Ytter Y. AGA Clinical Practice Guideline on Systemic Therapy for Hepatocellular Carcinoma. Gastroenterology. 2022 Mar;162(3):920-934. doi: 10.1053/j.gastro.2021.12.276. PMID 35210014
- [Result] Kudo M, Kawamura Y, Hasegawa K, Tateishi R, Kariyama K, Shiina S, Toyoda H, Imai Y, Hiraoka A, Ikeda M, Izumi N, Moriguchi M, Ogasawara S, Minami Y, Ueshima K, Murakami T, Miyayama S, Nakashima O, Yano H, Sakamoto M, Hatano E, Shimada M, Kokudo N, Mochida S, Takehara T. Management of Hepatocellular Carcinoma in Japan: JSH Consensus Statements and Recommendations 2021 Update. Liver Cancer. 2021 Jun;10(3):181-223. doi: 10.1159/000514174. Epub 2021 May 19. PMID 34239808
- [Result] Ruarus AH, Barabasch A, Catalano O, Leen E, Narayanan G, Nilsson A, Padia SA, Wiggermann P, Scheffer HJ, Meijerink MR. Irreversible Electroporation for Hepatic Tumors: Protocol Standardization Using the Modified Delphi Technique. J Vasc Interv Radiol. 2020 Nov;31(11):1765-1771.e15. doi: 10.1016/j.jvir.2020.02.030. Epub 2020 Sep 22. PMID 32978054
- [Result] Freeman E, Cheung W, Ferdousi S, Kavnoudias H, Majeed A, Kemp W, Roberts SK. Irreversible electroporation versus radiofrequency ablation for hepatocellular carcinoma: a single centre propensity-matched comparison. Scand J Gastroenterol. 2021 Aug;56(8):942-947. doi: 10.1080/00365521.2021.1930145. Epub 2021 May 30. PMID 34057003
- [Derived] Cheng C, Xu M, Pan J, Chen Q, Li K, Xu D, Jing X, Lu Q, Yang H, Zhao Q, Deng Z, Jiang T. A multicenter, randomized, parallel-controlled clinical trial protocol to evaluate the safety and efficacy of irreversible electroporation compared with radiofrequency ablation for the treatment of small hepatocellular carcinoma. World J Surg Oncol. 2024 Dec 20;22(1):332. doi: 10.1186/s12957-024-03614-z. PMID 39707376